CLINICAL TRIAL: NCT06537674
Title: An Exploratory Clinical Study of the PRO of Pyrotinib Combined With Trastuzumab Subcutaneously Compared Intravenous Administration in the Treatment of HER2-positive Early Breast Cancer
Brief Title: Pyrotinib Combined With Trastuzumab Subcutaneously Compared Intravenous Administration in the Treatment of HER2-positive Early Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: OBU-BC-II-184
Record Dates: First submitted 2024-07-24; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: HER2+ Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: The patient received six cycles of neoadjuvant therapy (pyrotinib and trastuzumab purplitol and platinum-based drugs) and underwent radical mastectomy (breast-conserving surgery or total mastectomy) after treatment. After the operation, the doctor will give the corresponding treatment according to the results of the postoperative medical examination
  Interventions: Drug: Trastuzumab intravenous drip/Trastuzumab Subcutaneous Injection
- Group B: The patient went on to complete six cycles of neoadjuvant therapy (pyrotinib and trastuzumab) and underwent radical mastectomy (breast-conserving surgery or total mastectomy) after treatment. After the operation, the doctor will give the corresponding treatment according to the results of the postoperative medical examination
  Interventions: Drug: Trastuzumab intravenous drip/Trastuzumab Subcutaneous Injection

INTERVENTIONS:
Drug: Trastuzumab intravenous drip/Trastuzumab Subcutaneous Injection — Group A is Trastuzumab intravenous drip,Group B is Trastuzumab Subcutaneous Injection

SUMMARY:
This study evaluated the clinical benefits of intravenous administration of pyrotinib combined with trastuzumab subcutaneous preparation by comparing the efficacy and quality of life of intravenous administration in the treatment of HER2-positive early breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥18 years and ≤75 years who are newly treated for breast cancer;
2. Pathological examination confirmed HER2 positive (immunohistochemical staining ICH+++ or ICH++ and FISH positive);
3. Patients with invasive breast cancer diagnosed histologically plus imaging as early (T1c-3, N0-1, M0) or locally advanced (T2-3, N2, or N3, M0);
4. ECOG score 0-1;
5. Plan to undergo the final surgical removal of breast cancer, i.e. breast-conserving surgery or total mastectomy, sentinel lymph node (SN) biopsy or axillary lymph node dissection (ALND);
6. If the major organs function normally, the following criteria are met:

(1) The standard of blood routine examination should meet: ANC ≥1.5×109/L; PLT ≥90×109/L; Hb ≥90g/L; (2) Biochemical examination should meet the following criteria: TBIL≤ upper limit of normal value (ULN); ALT and AST≤1.5 times the upper limit of normal (ULN); Alkaline phosphatase ≤2.5 times the upper limit of normal (ULN); BUN and Cr≤1.5×ULN and creatinine clearance ≥50 mL/min (Cockcroft-Gault formula); (3) Color Doppler ultrasonography and echocardiography: left ventricular ejection fraction (LVEF≥55%); (4) Fridericia calibrated QT interval (QTcF) for 18-lead ECG <470 ms; 7. For female patients who are not menopausal or have not been surgically sterilized, they should consent to abstinence or use an effective contraceptive method during treatment and for at least 7 months after the last dose in the study treatment.

8. Volunteer to join the study and sign the informed consent.

Exclusion Criteria:

1. Known allergic history of the drug components of this protocol;
2. Previously received antitumor therapy or radiation therapy for any malignant tumor (except for cured cervical carcinoma in situ and basal cell carcinoma);
3. Has undergone major non-breast cancer related surgery within 4 weeks, or has not fully recovered from such surgery;
4. Stage IV (metastatic) breast cancer patients;
5. Inability to swallow, intestinal obstruction, or other factors affecting the administration and absorption of the drug;
6. Serious heart disease or discomfort that cannot be treated;
7. Suffering from mental illness or psychotropic substance abuse, unable to cooperate;
8. Pregnant or lactating women;
9. Patients with severe liver and kidney function diseases and blood system diseases;
10. Those who were not considered suitable for inclusion by the researchers included: history of drug abuse, history of use of blood products, anticoagulant drugs and immunological drugs within the past year; Poor compliance and refusal to cooperate with treatment

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: HER2-positive early stage breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-C30 scale score | through study completion, an average of 1 year
  PRO scale scores between two groups collected at different time points

SECONDARY OUTCOMES:
tpCR | 1-2 weeks after surgery
  total pathological complete response